CLINICAL TRIAL: NCT06001918
Title: Randomized Controlled Clinical Trial (RCT) of the Nectero EAST System for Small to Mid-Sized Abdominal Aortic Aneurysms (AAA) StaBiLization: Evaluation of Efficacy.
Brief Title: Nectero EAST System Clinical Study
Acronym: stAAAble
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nectero Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAST002
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled trial comparing the efficacy of the treatment arm to the control arm.
Who Masked: Outcomes Assessor
Masking Description: For this trial, neither the patient nor investigator will be blinded to the study group assignment. However, members of the Sponsor, the CT core laboratory and the various committees reviewing subject data, such as the Clinical Events Committee (CEC), will be blinded to the randomization and assignment arm for an individual subject under review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Participants assigned to the treatment arm will undergo an endovascular procedure using the Nectero EAST System to deliver the Stabilizer Infusion Solution directly inside the aneurysm. This is a one-time local delivery of the product. Following treatment, surveillance of their AAA will be conducted using CT scans at 6 months, 12 months, 18 months, 24 months, and annually for 5 years.
  Intervention: Drug: Stabilizer
  Interventions: Drug: Nectero EAST System
- Control Arm (No Intervention): Participants assigned to the control arm will undergo surveillance of their AAA using CT scans at 6 months, 12 months, 18 months, 24 months, and annually for 5 years.

INTERVENTIONS:
Drug: Nectero EAST System — Treated subjects will undergo an endovascular procedure with the Nectero EAST system and receive the Stabilizer Infusion Solution (drug) within 30 days of the study eligibility by CT scan as a one-time local delivery of the drug.
  Arms: Treatment Arm

SUMMARY:
The purpose of this randomized clinical trial is to treat patients with small to mid-sized abdominal aortic aneurysms (AAA), maximum diameter of 3.5 cm to 5.0 cm, using a locally delivered, single-dose endovascular treatment. The main question the study aims to answer is to demonstrate efficacy of the product for stabilization of these small to mid-sized AAA.The study will compare the treatment group to the typical standard of care for these patients, surveillance. All subjects will be followed at designated intervals at 30/60 days, 6, 12, 18 and 24 months with continued follow-up annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥21 to ≤85 years of age. Females must be of non-childbearing potential (menopause or sterilization).
2. Subject understands the purpose of the trial, agrees to voluntarily participate in the trial, signs the informed consent and is willing to complete the follow-up according to the requirements of the protocol.
3. Infrarenal atherosclerotic fusiform abdominal aortic aneurysm from 3.5 cm to 5.0 cm (male) and 3.5 cm to 4.5 cm (female).
4. Infrarenal aortic neck ≥ 15 mm in length and ≤ 29 mm in diameter.
5. Overall AAA treatment length (distal renal to distal inferior margin of the aneurysm) not to exceed 130 mm.
6. Iliac and femoral artery access, vessel size and morphology allow endovascular access of 14F (or larger) introducer sheaths and catheters.
7. Subject meets American Society of Anesthesiology (ASA) grade 1 through 3 criteria, inclusive.
8. Subject has > three-year life expectancy.
9. Subject is able and willing to comply with all required follow-up clinic visits including CT scans (pre-randomization, 6, 12, 18, 24 months and annually up to 5 years) and blood draws.

Exclusion Criteria:

1. Subject has an acutely ruptured, leaking, dissecting or emergent aneurysm.
2. Subject has a symptomatic infrarenal abdominal aortic aneurysm.
3. Subject has a mycotic or infected aneurysm.
4. Subject has current vascular injury due to trauma.
5. Subject's aneurysm is thoracic, suprarenal or juxtarenal.
6. Previous surgical or endovascular aneurysm repair for abdominal aortic aneurysm.
7. Subject has anatomy of diffuse, ulcerated, or extensive (shaggy) thrombus in the neck of the AAA, that in the opinion of the vascular surgeon/investigator, could result in embolization of the thrombus.
8. Subject has anatomy of calcification, and/or plaque within the ilio-femoral arteries or severe infrarenal neck angulation that may compromise or does not allow delivery of the Introducer Sheath or the delivery catheter of the Nectero EAST System.
9. Subject has had a myocardial infarction within six (6) months prior to enrollment or elevated CK enzymes or troponin indicative of an evolving MI prior to procedure.
10. Subject has current angina, unstable angina, or other active cardiac condition such as congestive heart failure III and IV, atrial arrhythmia, ventricular arrhythmia, or valvular disease, requiring intervention.
11. Subject has undergone other major surgery within the 30 days prior to enrollment.
12. Subjects with any transient ischemic attack (TIA) or ischemic stroke within 3 months.
13. Known allergy to contrast material that cannot be adequately premedicated, delivery system materials (i.e., nylon, polyurethane) and/or pentagalloylglucose (PGG).
14. Subject is morbidly obese or has other clinical conditions that severely inhibit X-ray visualization of the aorta.
15. Subject has connective tissue/collagen disorder (e.g., Marfan syndrome, vascular Ehlers-Danlos Syndrome, Loeys-Dietz Syndrome, Eaton Syndrome, Bessel-Hagen disease, etc.).
16. Known contraindication to undergoing angiography or receiving systemic anticoagulation during the procedure.
17. Subject has active systemic infection.
18. Subject is participating in another research trial that could interfere with the results of the trial (e.g., drug trial).
19. Subject has other medical, social, or psychological problems that, in the opinion of the investigator, preclude them from participation in the trial and to undergo the procedures and evaluations pre- and post-treatment.
20. Subject has dialysis dependent renal failure or baseline serum creatinine level >2.5mg/dL or eGFR < 45 mL/min/1.73m2.
21. Subjects with aminotransferase (ALT and/or AST) which is ≥1.5x upper limit of normal (ULN) or TB that is our of normal range for the evaluating laboratory.
22. Subjects that may not tolerate the lowering of their systolic blood pressure to approximately 100mmHg, should not be considered for this study or treated using the Nectero EAST System.
23. Subjects that may not be able to tolerate transient occlusion of the aorta should not be considered for this study.
24. Subjects with saccular AAA.
25. Subjects with rapidly expanding AAA (previous diameter increases of ≥0.5 cm in 6-months or ≥1 cm in 1 year) as these should be evaluated for immediate repair.
26. Subjects who are not suitable for the Nectero EAST System treatment, as determined by the investigator.
27. Subjects with INR out of normal range for the evaluating laboratory for a subject not on anti-coagulant therapy; or INR >3 for a subject on anti-coagulant therapy.
28. Subjects with active/acute or a history of unstable chronic liver disease or current liver disease including but not limited to liver transplant, known genetic disorders such as Gilbert syndrome or other liver diseases.
29. Subjects with cirrhosis (e.g., known history or new clinical diagnosis by elastography with a fibrosis score of F3 or F4 and/or steatosis grade of S3).
30. Subjects with uncontrolled alcohol use disorder or current alcohol use putting them at risk of liver disease: including consumption of above one standard drink per day for women and two standard drinks per day for men.
31. Subjects with known right-sided heart failure or pathologically dilated inferior vena cava or hepatic veins indicative of congestive hepatopathy.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 24 months
  The primary endpoint is the composite of all AAA-related death, rupture and repair (open-surgical, EVAR, or clinically indicated for repair as adjudicated by a committee of clinical experts blinded to the assigned arm).

SECONDARY OUTCOMES:
Growth | 24 months
  The growth over time in aneurysm diameter based on CT core laboratory readings.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, MD, Principal Investigator — Vanderbilt University Medical Center; Grace Wang, MD, Principal Investigator — University of Pennsylvania
Locations (39):
- United States (37):
  - Honor Health Scottsdale Shea Medical Center, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Prime Vascular Institute, Delray Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - MaineMed Vascular Surgery, Scarborough, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Beaumont Health, Royal Oak, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Rochester, Rochester, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Ohio Health Riverside, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Portland VA Medical Center, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Clinical Research Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - North Central Heart - A Division of Avera Heart Hospital, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Healthcare, Houston, Texas
  - Baylor Scott & White Medical Center, Plano, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Medical Campus Inova Health Systems, Fairfax, Virginia
  - University of Washington at Harborview Medical Center, Seattle, Washington
  - Bellin Memorial Hospital, Green Bay, Wisconsin
- Prince of Wales Private Hospital- POW Vascular Institute, Randwick, New South Wales, Australia
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- [Background] Cheng SWK, Eagleton M, Echeverri S, Munoz JG, Holden AH, Hill AA, Krievins D, Ramaiah V. A pilot study to evaluate a novel localized treatment to stabilize small- to medium-sized infrarenal abdominal aortic aneurysms. J Vasc Surg. 2023 Oct;78(4):929-935.e1. doi: 10.1016/j.jvs.2023.05.056. Epub 2023 Jun 15. PMID 37330148
- See also: J Vasc Surg. Pilot Study — https://pubmed.ncbi.nlm.nih.gov/37330148/